CLINICAL TRIAL: NCT00871442
Title: Parturient Controlled Epidural Analgesia (PCEA) With or Without a Basal Infusion for Early Labor
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: would not substantially add to existing contributions in the literature
Sponsor: Neil Roy Connelly, MD (Other)
Responsible Party: Sponsor-Investigator, Neil Roy Connelly, MD, Anesthesiologist, Baystate Medical Center
Organization: Baystate Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB09-017
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2009-07

CONDITIONS: Labor Pain
Keywords: PCEA; labor and delivery; pain; epidural; anesthesia; pregnant women
MeSH Terms: conditions — Labor Pain; Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Basal Infusion (Active Comparator): PCEA solution: Bupivacaine 0.0625% with fentanyl 2 mcg/ml
  Group 1: Basal Infusion: 0 ml/hr; Bolus 10 ml q 30min prn (10ml demand dose with 30min lockout)
  Interventions: Other: No Basal Infusion; Drug: PCEA solution (bupivacaine and fentanyl)
- Basal Infusion (Active Comparator): PCEA solution: Bupivacaine 0.0625% with fentanyl 2 mcg/ml
  Group 2: Basal Infusion: 10 ml/hr; Bolus 5 ml q 30min prn (5ml demand dose with 30min lockout)
  Interventions: Other: Basal infusion; Drug: PCEA solution (bupivacaine and fentanyl)

INTERVENTIONS:
Other: No Basal Infusion — Group 1: Basal Infusion: 0 ml/hr; Bolus 10 ml q 30min prn (10ml demand dose with 30min lockout)
  Other Names: epidural infusion; bupivicaine; patient controlled epidural anesthesia (PCEA); PCEA pump settings
  Arms: No Basal Infusion
Other: Basal infusion — Group 2 Basal Infusion: 0 ml/hr; Bolus 10 ml q 30min prn (10ml demand dose with 30min lockout)
  Other Names: epidural infusion; bupivicaine; patient controlled epidural anesthesia (PCEA); PCEA pump settings
  Arms: Basal Infusion
Drug: PCEA solution (bupivacaine and fentanyl) — PCEA solution: Bupivacaine 0.0625% with fentanyl 2 mcg/ml

SUMMARY:
Patient Controlled Epidural Analgesia is a widely used and effective means of adult pain management. However, Parturient Controlled Epidural Analgesia (PCEA) is a relatively new approach to pain control for the women in labor. With the recent acquisition of new PCEA technology at Baystate Medical Center it is now possible to make this patient controlled technology available on the Labor and Delivery unit. This study is designed to determine whether there is a difference in analgesia, side effects, or analgesic duration in patients who receive a bupivacaine and fentanyl PCEA for management of labor pain. The present study hypothesizes that an analgesic protocol that includes a basal infusion rate in addition to a bolus dose controlled by the patient will have a longer analgesic duration than a pump protocol that does not have a basal infusion added to a bolus dose controlled by the patient.

Methods:The study population will consist of 100 adult obstetrical patients greater than 36 weeks gestation who request labor analgesia. Patients greater than 5 cm cervical dilation, patients who have received intravenous opioid agonists, or patients with a contraindication to fentanyl will be excluded. Patients with pre-eclampsia are also excluded.

One of the following PCEA treatment protocols will be started in a randomized, double blind fashion.PCEA solution: Bupivacaine 0.0625% with fentanyl 2 mcg/ml Group 1: Basal Infusion: 0 ml/hr; Bolus 10 ml q 30min prn (10ml demand dose with 30min lockout) Group 2: Basal Infusion: 10 ml/h; Bolus 5 ml q 30min prn (5ml demand dose with 30min lockout) If the patient does not obtain relief within 30 minutes, the epidural catheter will be dosed with a local anesthetic and the study will be concluded. The patients without pain relief within 30 minutes are considered to have failed epidurals and are dropped from the study and the analysis. Following achievement of satisfactory analgesia, the patient will be evaluated every 30 minutes until they request additional analgesics. The study will "end" at this point, and the patient will be treated at the discretion of the anesthesiologist.

DETAILED DESCRIPTION:
Patient Controlled Epidural Analgesia is a widely used and effective means of adult pain management. However, Parturient Controlled Epidural Analgesia (PCEA) is a relatively new approach to pain control for the women in labor. With the recent acquisition of new PCEA technology at Baystate Medical Center it is now possible to make this patient controlled technology available on the Labor and Delivery unit. Several studies have been conducted to evaluate the effects of Parturient Controlled Epidural Analgesia on different outcomes ranging from the dose of local anesthetic used, incidence of motor block, quality of analgesia, obstetric and safety outcomes, and number of patients who received anesthetic interventions.

We have previously shown that epidural fentanyl (given in a 10 ml volume) is a useful means of achieving analgesia in laboring patients receiving epidural analgesia. Furthermore, we have shown that adding a bupivacaine and fentanyl infusion increases the analgesic period. This increased analgesic duration was achieved without any clinically detectable motor block. This study is designed to determine whether there is a difference in analgesia, side effects, or analgesic duration in patients who receive a bupivacaine and fentanyl PCEA for management of labor pain. The present study hypothesizes that an analgesic protocol that includes a basal infusion rate in addition to a bolus dose controlled by the patient will have a longer analgesic duration than a pump protocol that does not have a basal infusion added to a bolus dose controlled by the patient.

Methods:

The study population will consist of 100 adult obstetrical patients greater than 36 weeks gestation who request labor analgesia. Patients greater than 5 cm cervical dilation, patients who have received intravenous opioid agonists, or patients with a contraindication to fentanyl will be excluded. Patients with pre-eclampsia are also excluded.

The screening process occurs when the patient requests labor analgesia. The study is then explained to the patient as well as the option of receiving labor analgesia without participating in the study protocol. The epidural catheters will be placed in the usual fashion in the L2-3 interspace. The catheter will be injected with 3ml lidocaine 1.5% with epinephrine 1:200,000 "test dose" (as is the usual practice at Baystate following insertion of all epidural catheters) to rule out placement of an intravenous catheter. All catheters will be placed in 5 cm. Following customary test dosing, patients will be given Fentanyl 100 mcg in 10 ml volume. After the woman is comfortable from the epidural, we will again approach the patient. If the patient then agrees to participate in the study and signs the consent form, study procedures are initiated.

One of the following PCEA treatment protocols will be started in a randomized, double blind fashion. A random number table for 60 patients is generated in Excel using the Randbetween function. This function randomly generates 60 numbers either 1 or 2. When a series is generated that contains 30 1's and 30 2's, this series is selected as the random code for the study. A patient is assigned to group 1 or 2 based on the next available number. This patients name is then entered next to this number on the rand code table.

PCEA solution: Bupivacaine 0.0625% with fentanyl 2 mcg/ml

Group 1: Basal Infusion: 0 ml/hr; Bolus 10 ml q 30min prn (10ml demand dose with 30min lockout) Group 2: Basal Infusion: 10 ml/h; Bolus 5 ml q 30min prn (5ml demand dose with 30min lockout)

The pump will be programmed by one investigator while evaluations will be done by another investigator who is unaware of the PCEA protocol.

If the patient does not obtain relief within 30 minutes, the epidural catheter will be dosed with a local anesthetic and the study will be concluded. The patients without pain relief within 30 minutes are considered to have failed epidurals and are dropped from the study and the analysis. Following achievement of satisfactory analgesia, the patient will be evaluated every 30 minutes until they request additional analgesics. The study will "end" at this point, and the patient will be treated at the discretion of the anesthesiologist.

Method of delivery, need for instrumented delivery, time of delivery, and neonatal APGAR scores will be recorded.

The level of discomfort, presence of side effects (motor block, sedation, pruritis, and hypotension) will be evaluated at baseline, 10, 20, 30 minutes and every 30 minutes thereafter. Pain will be evaluated using a 100-mm visual analogue scale (VAS) with 0 representing no pain and 100 representing the worst possible pain. We will track several PCEA parameters including volumes infused till study termination, Bolus Demands, Bolus Deliveries, time to first bolus etc.

All other aspects of the patients' care will conform to usual standards.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of 100 adult obstetrical patients greater than 36 weeks gestation who request labor analgesia.

Exclusion Criteria:

* Patients greater than 5 cm cervical dilation,
* Patients who have received intravenous opioid agonists,
* Patients with a contraindication to fentanyl, OR
* Patients with pre-eclampsia are also excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Analgesic duration | request for analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Neil Roy Connelly, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States